CLINICAL TRIAL: NCT01082770
Title: A Randomised Controlled Trial Comparing Bacteraemia Rates in Closed Luer Lock Access Devices(TEGO) With Standard Devices in the Outpatient Haemodialysis Population
Brief Title: Randomised Controlled Trial of Needle Free Access Devices in Preventing Hemodialysis Blood Stream Infection
Acronym: TEGO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beaumont Hospital (Other)
Responsible Party: Professor Peter Conlon, Beaumont Hospital, Dublin 9, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TEGOIRL
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-01

CONDITIONS: Hemodialysis Catheter Blood Stream Infection; Central Line Infection; Dialysis Line Thrombosis
MeSH Terms: interventions — Reference Standards

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TEGO (Active Comparator): TEGO needle free access devices will be used in patients randomised to this arm
  Interventions: Device: TEGO
- Control (Placebo Comparator): Patients will continue to receive current standard of practice, ie a 'bung' cap at the end of the hemodialysis line
  Interventions: Device: Standard

INTERVENTIONS:
Device: TEGO — A bung that can be attached to the end of dialysis lines that can be directly attached to the dialysis machine with minimal handling
  Arms: TEGO
Device: Standard — Patients in this group will have a normal 'bung' placed at the end of their dialysis line, which will need to be removed by nursing staff prior to initiation of dialysis
  Arms: Control

SUMMARY:
This study will be a randomised controlled trial examining whether a new type of needle free access device(TEGO) is associated with less episodes of infection of dialysis lines, when compared to the current gold standard.

The investigators hypothesise that there will be less handling of the dialysis line by nursing staff and thus this will lead to lower rates of infection. The investigators will also assess whether these access devices lead to alterations in catheter blood flow rates when compared to the current gold standard.

DETAILED DESCRIPTION:
Introduction

Infection is an important cause of morbidity and mortality in patients with ESKD. Examining the USRDS database, it is the second leading cause of death in these patients . Several studies in the past number of years have highlighted permanent vascular access devices as independent risk factors for the development of sepsis .

Approximately 50% of haemodialysis patients in Beaumont Hospital use permanent central catheters, often while awaiting alternative vascular access, such as arterio-venous fistulae or when other avenues of vascular access have been exhausted. International data has shown that patients with permanent vascular access devices have 50% higher infection rates compared to those with a native fistula .

Permanent central venous catheters used in haemodialysis are tunnelled cuffed dual lumen catheters usually composed of silicone or polyurethane materials. These are usually placed in the right internal jugular vein. Tunnelled haemodialysis catheters are placed in the radiology department under fluoroscopic guidance.

The presence of catheter related bacteraemia is often treated with intravenous antibiotics such as vancomycin or gentamycin, however a study of 100 haemodialysis patients in Ann Int Med in 1997 has shown that attempts to treat bacteraemia without removal of the catheter usually fail . In such cases, removal of the catheter and insertion of another at either the same or another site is necessary.

Methods of reducing catheter related bacteraemia such as intensive hygiene education, the use of cuffed catheters and the use of prophylactic antibiotic therapy have all been employed, however with limited success

It is hypothesised that repeated opening and handling of the catheter increase the risk of bacteraemia, and so a closed luer lock access device would reduce bacteraemia rates.

Several studies have shown reductions in catheter bacteraemia when closed luer lock devices were used in an ITU setting . Little data exists on infection rates in out patient haemodialysis setting.

A recent study in NDT examining the blood flow resistance of these closed lock access devices show values within safe ranges, suggesting that these devices can safely be used in the out patient haemodialysis setting.

Objective

To identify if a closed luer lock access devices can result in lower rates of bacteraemia and/or sepsis in patients receiving haemodialysis through a permanent vascular catheter when compared to current practise methods.

Primary End Points:

Episodes of bacteraemia or line sepsis requiring antibiotic therapy. Bacteraemia will be defined as positive blood culture specimen.

Bacteraemia will be defined as any episode of temperature > 38º or <36º will be an indication to perform blood cultures, as will cellulitis around catheter sites. A positive blood culture result will be labelled a catheter related bacteraemia if no other obvious source of infection is noted. The physician attending the patient for the above reasons will perform a full physical exam and request an MSU if possible from all patients seen to aid accuracy of results.

Secondary End Points:

Renal blood flow rates in the closed luer lock devices when compared to the standard access devices.

Renal blood flow rates will be recorded by the haemodialysis nursing staff at each dialysis session.

Incidence of line obstruction requiring thrombolytic therapy in the closed luer lock device when compared to standard devices.

Incidence of thrombolytic use will be recorded by the attending haemodialysis nurse.

This study hypothesises that closed luer lock access devices will lead to significantly reduced rates of catheter related bacteraemia, and thus reduced patient morbidity and mortality. It is also hypothesised that renal blood flow rates will be higher in the TEGO study group

Methods

This study will be designed as a one centre prospective randomised case control study, taking place in Beaumont Hospital in St Martin's dialysis wards and St Peter's dialysis ward over a twelve month period.

It shall run from December 2009 to December 2010, with the aim of recruiting 100 patients for the study, 50 patients in the control group and 50 in the treatment group. All patients will receive fully informed written consent prior to entering the trial.

Patients will be randomised into both groups using sequentially numbered, opaque sealed envelopes.

Patients may withdraw from the study at any time with no implications for his/her haemodialysis treatment regime. Patients who undergo transplantation during the trial will be removed from the study at that time, and data collected up to the time of transplantation will be incorporated into the study.

Inclusion criteria Patients recruited will be over 18 and have been on haemodialysis for greater than one month, have permanent cuffed vascular access lines in place and will be receiving haemodialysis through these lines three times per week.

Patients will not have had a documented episode of bacteraemia or sepsis for greater than 4 weeks, and will not be using antibiotic coated dialysis lines.

Exclusion criteria Patients with immunosuppressive illnesses such as HIV, cancer or patients who regularly use glucocorticoids.

Study group Patients in the study group will use TEGO® devices on both access ports, which will be changed after one week or 25 uses. This device which costs €2.30, and will be supplied gratis by Fannin Ltd Dublin and ICU Medical Inc, San Clemente USA.

TEGO® devices will be accessed by the haemodialysis nursing staff using aseptic technique.

Control group Patients in the control group will continue to receive haemodialysis using the current standard of care protocol.

Data Collection Bacteraemia rates from each group will be recorded by the haemodialysis nursing staff and subsequently will be inputted into a Microsoft Excel spreadsheet. Further analysis including comparison of both patient groups will take place using SPSS software. Data will only be stored on a hospital server, and will only be accessible by members of the research team.

The power of the study will be calculated using Fisher's combined probability test, where Test Ho: p1=p2, where p1 is in proportion in population 1 and p2 is in proportion in population 2. Assumptions:

Alpha = 0.0500 (two sided) Power = 0.8000 P1 = 0.17 P2 = 0.000 N2/N1 = 1.00

Estimated sample sizes

N1 = 53 N2 = 53

Subsequent data analysis will include comparison of outcomes using a student's t test and subsequent formation of Kaplan Meier curves.

ELIGIBILITY:
Inclusion Criteria:

* Patients recruited will be over 18 and have been on haemodialysis for greater than one month, have permanent cuffed vascular access lines in place and will be receiving haemodialysis through these lines three times per week.
* Patients will not have had a documented episode of bacteraemia or sepsis for greater than 4 weeks, and will not be using antibiotic coated dialysis lines.

Exclusion Criteria:

* Patients with immunosuppressive illnesses such as HIV, cancer or patients who regularly use glucocorticoids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Bacteraemia rates in the needle free access devices(TEGO) when compared to current practice | 1 year
  New needle free access devices will be compared to current 'bung' devices. Patients will be randomly assigned to both groups, and rates of bacteraemia will be compared between both groups

SECONDARY OUTCOMES:
Catheter blood flow rates in study device compared to control | 1 year
  Safety of new TEGO, needle free access device will be assessed by measuring the catheter blood flow rates in the study group compared to the control group
Rates of line thrombosis in study group compared to control group | 1 year
  Rates of line thrombosis requiring t-PA administration will be compared in the study group and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Peter Conlon, MD, Study Chair — Beaumont Hospital Dublin
Locations (1):
- Beaumont Hospital, Dublin, Dublin, Ireland